CLINICAL TRIAL: NCT02404012
Title: Comparison of Iron Supplement Formulations to Improve Iron Status Following Roux-en-Y and Sleeve Gastrectomy Bariatric Surgery
Brief Title: Iron Supplement to Improve Iron Status Following Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nana Gletsu Miller, Assitant Prof. Nutrition Sciences, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB1410015305
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Anemia, Iron Deficiency
Keywords: iron deficiency; sleeve gastrectomy; gastric bypass; bariatric surgery
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous sulfate (Active Comparator): Ferrous sulfate 65 mg. t.i.d is the standard of care for oral supplementation for iron deficiency
  Interventions: Dietary Supplement: Oral iron supplementation
- AspironTM 65 mg t.i.d. (Experimental): AspironTM, an organic formulation of iron, is the experimental treatment for oral supplementation of iron deficiency
  Interventions: Dietary Supplement: Oral iron supplementation

INTERVENTIONS:
Dietary Supplement: Oral iron supplementation — Participants will be provided supplementation for 8 weeks

SUMMARY:
There is a high prevalence of iron deficiency in patients who undergo bariatric surgery and effective therapies are lacking. Thus, there is a critical need for an effective, non-invasive, and inexpensive form of iron supplementation to treat iron deficiency and improve tolerance, the associated cognitive symptoms, and quality of life in the bariatric surgery patient population. Often, patients do not participate in bariatric programs, are not compliant, and/or are lost to follow-up. If there is a more effective and evidence-based guideline for repletion of iron deficiency, patients are more likely to be compliant. Therefore, in a randomized controlled study, the investigators propose to test the effectiveness of various iron formulations versus ferrous sulfate, which is the standard of care, for oral iron supplementation of iron deficient patients who have had RYGB or SG bariatric surgery. By randomizing patients into the two groups, the investigators will be able to determine the most effective regimen to improve blood biomarkers of iron status, cognitive function, and quality of life. Other outcomes will include adverse effects and compliance to the supplementation. The investigators will also analyze three-day food records to determine the contribution of dietary factors to changes in iron status. To test for improvement of iron status, serial blood draws will be performed during a time period of ~10 weeks. Serial blood draws from iron deficient patients have routinely been performed in past studies and have not been found to be harmful. Because this is a relatively short study (10 weeks), subjects will be able to recover quickly from the blood loss during the study. The investigators expect to find that iron supplementation with organic formulations of iron will be as effective than ferrous sulfate for repletion of iron deficiency, and they will be better tolerated. This project will address a significant health issue in individuals who have had bariatric surgery, which is a growing population in the United States. It is estimated that almost 1.5 million individuals have undergone bariatric surgery since the year 1990.

DETAILED DESCRIPTION:
Objectives:

1. To determine the most effective oral iron supplementation regimen for repletion of iron deficiency in patients who have had gastric bypass or sleeve gastrectomy. In iron deficient patients, two supplement regimens will be compared:

   1. Ferrous sulfate 65 mg t.i.d. (standard of care / control), which is elemental iron
   2. AspironTM, which is an organic formulation of iron

   Primary outcomes will be reference indices of iron status:
   * Ferritin, TIBC, sTfR, and sTfR:ferritin ratio
   * Secondary outcomes will be:
   * measures of anemia, determined by blood hemoglobin concentrations
   * measures of cognitive function via several computerized tests on working memory, sustained attention, and spatial memory
   * fatigue by Multidimensional Fatigue Inventory questionnaire
   * Quality of life by SF-36 Survey

   Safety outcomes will be:

   • adverse events, compliance, measures of iron toxicity, and liver enzymes
2. In the same subjects undergoing iron supplementation described in Aim 1, to determine the contribution of dietary factors (including heme and non-heme iron intake, and intake of enhancers and inhibitors of iron absorption) to changes in iron status.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a history of RYGB or SG weight loss surgery at least 6 months ago
* Subject meets at least 2 of the 4 previously mentioned conditions classifying them as iron deficient
* Subject is female
* Subject is at least 18 but not more than 65 years of age (post-menopausal status is an exclusion criteria)
* Subject has signed an informed consent.

Exclusion Criteria:

* Subject is pregnant
* Subject has history of surgical revision or conversion of bariatric procedure
* Subject is under a treatment regimen that requires iron supplementation greater than standard of care
* Subject has had parenteral iron less than one month before screening visit
* Subject has extremely heavy menstruation
* Subject has a history of hospitalization for acute illness in the previous 3 months
* Subject has current active malignant neoplasm; or history of malignancy other than localized basal cell cancer of skin during previous 5 years
* Subject has gastrointestinal disease that involve increased inflammation or blood loss (e.g. Crohn's disease, Ulcerative colitis)
* Subject is post-menopausal
* Subject has severe anemia, with a hemoglobin > 7.0 g/dL (subjects will be notified of their results)
* Subject is taking an erythropoietin stimulating medication or is on hemodialysis.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-11; Primary Completion 2019-12 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Iron status | 8 weeks
  Ferritin, TIBC, sTfR

SECONDARY OUTCOMES:
Anemia assessed by Hemoglobin concentrations | 8 weeks

OTHER OUTCOMES:
Safety outcomes assessed by adverse events, compliance | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- Available data/document: Website — https://ngletsum.wixsite.com/nito